CLINICAL TRIAL: NCT05304676
Title: Additional Effects of Kinesio Tape and Neuromuscular Electrical Stimulation on the Hand Activity in Hemiplegic Cerebral Palsy
Brief Title: Additional Effects of Kinesiotape and Neuromuscular Electrical Stimulation on the Hand Activity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01039 Umair
Record Dates: First submitted 2022-01-21; First posted 2022-03-31 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KTT group (Experimental): This group will receive neurodevelopmental treatment along with kinesotape and neuromuscular electrical stimulation. Children will be treated for 3 days a week over 4 weeks.
  Interventions: Other: Experimental: KTT group
- Conventional treatment (Active Comparator): Group B will receive neurodevelopment treatment along with neuromuscular electrical stimulation.
  Interventions: Other: Active Comparator: conventional treatment

INTERVENTIONS:
Other: Experimental: KTT group — This group will receive neurodevelopmental treatment along with kinesotape and neuromuscular electrical stimulation
  Arms: KTT group
Other: Active Comparator: conventional treatment — Group B will receive neurodevelopment treatment along with neuromuscular electrical stimulation.
  Arms: Conventional treatment

SUMMARY:
Children with cerebral palsy (CP) manifest several developmental disorders of movement and posture. CP children have functional limitations so this study investigates the additional effects of kinesio taping and neuromuscular electrical stimulation on hands joint range of motion, muscle tone and functional ability in children with hemiplegic cerebral palsy

DETAILED DESCRIPTION:
Hemiplegia is a form of spastic Cerebral Palsy (CP) in which one arm and leg on either the right or left side of the body is affected. It is the most common syndrome in children born at term and is second in frequency only to spastic diplegia among preterm infants. Patients with spastic hemiplegia have unilateral prehensile dysfunction as a consequence of lesions in the sensorimotor cortex and corticospinal tract. The upper limb is usually more severely involved than lower one. This limit reaching, grasping and object manipulation, interfering also with exploration, play, self-care and other activities of daily living. It is the most common cause of severe physical disabilities in childhood, in which hemiplegia is accounted for 36% of children with cerebral palsy. Children with hemiplegic cerebral palsy usually have the independent walking ability and intellectual capacity to attend regular school. However, impaired hand function restricts their activity and participation in lifestyle, educational, leisure and later vocational roles. The most common postures of the upper extremity in children with cerebral palsy are shoulder internal rotation, elbow flexion, forearm pronation, wrist flexion, finger flexion and thumb in palm is a very common problem seen in children with cerebral palsy (CP) and its solution is difficult. The deformity is complex and can include: contracture of the thumb metacarpophalangeal joint or global instability; contractures of the intrinsic muscles and spasticity; extrinsic motor imbalance with over lengthening and/or weakness of the extensor pollicus longus, extensor pollicus brevis, and abductor pollicus longus; and contracture and/or weakness of the flexor pollicus longus. Thumb in palm deformity can cause restrictions in functional ability and prevent somatosensory input in these children. Kinesio taping (KT) is a relatively new therapeutic tool used in rehabilitation program of children with cerebral palsy, although it has been used for a long time in sport or orthopedic fields, and has been approved as a supplemental intervention for other functional impairments. Kinesio tape is a specialized elastic-like tape made of latex-free cotton fibers having no medication effect and designed to mimic the elasticity properties of the muscle, skin and fascia. By proper taping, the elasticity of the tape not only does not restrict the soft tissue, but also supports the weak muscles and creates a full ROM.(8) An adjunct therapy, which has gained increasing support for CP in the 1970s is neuromuscular electrical stimulation (NMES). With NMES, electrical stimulation of sufficient intensity generally to produce visible muscle contraction is applied at the muscle motor point. Several case studies have reported improvement in hand function

ELIGIBILITY:
Inclusion Criteria:

* • Age: 3 year to 15 year

  * Gender: Both Male and female.
  * Diagnosis with hemiplegic cerebral palsy
  * Refer for physiotherapy
  * Classified as Gross Motor Function Classification System level II, III
  * Ashworth grading: 1-3
  * Able to follow and accept verbal instruction and communication

Exclusion Criteria:

* Medical procedures likely to affect motor function such as botulinum toxin injection.
* Any kind of surgery.
* Mental retardation or learning disability.
* Any other abnormality and pathology condition.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Jebsen Hand Function Test | 4 weeks
  The Jebsen Hand Function Test (JHFT/JTT) was developed to provide a standardized and objective evaluation of fine and gross motor hand function using simulated activities of daily living. It consists of seven subsets which are writing, simulated page-turning, lifting small objects, simulated feeding, stacking, and lifting large, lightweight, and heavy objects.Total score is the sum of time taken for each sub-test, which are rounded to the nearest second. Shorter times indicate better performance.Change from Baseline hand functions to 4th Week
Minnesota Hand Skill Test | 4 Week
  The Minnesota Manual Dexterity test (MMDT) tool was developed to measure unilateral and bilateral gross and fine manual dexterity.his involved a series of displacement and turning of plastic or wooden cylinders to be placed in a series of matched holes. A log is maintained of the time taken for these steps.Change from Baseline manual ability and hand dexterity to 4 Week
Goniometer | 4Week
  Goniometer is used to measure range of motion of joints, following joints will be assessed shoulder, elbow, wrist. Change from Baseline manual ability and hand dexterity to 4 Week

SECONDARY OUTCOMES:
Manual Ability Classification System | 4Weeks
  This proposed new classiﬁcation, the Manual Ability Classiﬁcation System (MACS), is designed to classify how children with CP use their hands when handling objects in daily activities. MACS describes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life.Change from Baseline manual ability and hand dexterity to 4 Week
Gross Motor Function Classification System | 4Weeks
  The gross motor function of children and young people with cerebral palsy can be categorized into 5 different levels using a tool called the Gross Motor Function Classification System. Change from Baseline manual ability and hand dexterity to 4 Week

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah college of Rehabilitation and Allied Health sciences Islamabad
Locations (2):
- Pakistan (2):
  - National Institute of Rehabilitation and Medicine, Islamabad
  - Misbah Ghous, Rawalpindi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozer K, Chesher SP, Scheker LR. Neuromuscular electrical stimulation and dynamic bracing for the management of upper-extremity spasticity in children with cerebral palsy. Dev Med Child Neurol. 2006 Jul;48(7):559-63. doi: 10.1017/S0012162206001186. PMID 16780624
- [Background] Sankar C, Mundkur N. Cerebral palsy-definition, classification, etiology and early diagnosis. Indian J Pediatr. 2005 Oct;72(10):865-8. doi: 10.1007/BF02731117. PMID 16272660
- [Background] Acıkbas E, Tarakcı D, Budak M. Comparison of the effects of Kinesio taping and neuromuscular electrical stimulation on hand extensors in children with cerebral palsy. Int J Ther Rehabil. 2020. https://doi.org/10.12968/ ijtr.2019.0053
- [Background] Kitai Y, Haginoya K, Hirai S, Ohmura K, Ogura K, Inui T, Endo W, Okubo Y, Anzai M, Takezawa Y, Arai H. Outcome of hemiplegic cerebral palsy born at term depends on its etiology. Brain Dev. 2016 Mar;38(3):267-73. doi: 10.1016/j.braindev.2015.09.007. Epub 2015 Oct 1. PMID 26428444